CLINICAL TRIAL: NCT06922877
Title: Diagnostic Accuracy of 3-dimensional Imaging Device on Polyps and Adenomas During Colonoscopy: a Single-center Randomized Controlled Trial
Brief Title: Diagnostic Accuracy of 3-dimensional Imaging Device on Polyps and Adenomas During Colonoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Zhiguo Liu, associate professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: KY20242178-F-1
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Polyps; Colorectal Adenomas
Keywords: three dimension imaging device; colorectal polyps; colorectal adenomas

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2D imaging arm (Active Comparator): participants will undergo polypectomy (CSP, CFP, or EMR) using 2D imaging colonoscope
  Interventions: Diagnostic Test: endoscopic evaluation of colorectal polyps and adenomas using 2D imaging colonoscope
- 3D imaging arm (Experimental): participants will undergo polypectomy (CSP, CFP, or EMR) using 3D imaging colonoscope
  Interventions: Diagnostic Test: endoscopic evaluation of colorectal polyps and adenomas using 3D imaging colonoscope

INTERVENTIONS:
Diagnostic Test: endoscopic evaluation of colorectal polyps and adenomas using 2D imaging colonoscope — endoscopic diagnostic evaluation of colorectal polyps and adenomas before polypectomy using 2D imaging colonoscope
  Arms: 2D imaging arm
Diagnostic Test: endoscopic evaluation of colorectal polyps and adenomas using 3D imaging colonoscope — endoscopic diagnostic evaluation of colorectal polyps and adenomas before polypectomy using 3D imaging colonoscope
  Arms: 3D imaging arm

SUMMARY:
The goal of this clinical trial is to learn if 3-dimensional (3D) imaging device works to correctly classify colon polyps and adenomas during colonoscopy to guide the selection of proper treatment procedures. It will also learn about the safety of 3-dimensional (3D) imaging device. The main questions it aims to answer are:

Does 3-dimensional (3D) imaging device improve the correct classification as well as size and depth evaluation of polyps and adenomas during colonoscopy using pathology as gold standard? What adverse events do participants experience during colonoscopy and polypectomy?

Researchers will compare 3-dimensional (3D) imaging device to traditional 2-dimensional (2D) imaging device to see if 3-dimensional (3D) imaging device works to improve classification and evaluation accuracy.

Participants will:

Undertake colonoscopy examination and polypectomy using 3-dimensional (3D) imaging device or 2-dimensional (2D) imaging device.

Be followed-up to 30 days to record potential colonoscopy-relevant adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years;
* Endoscopically diagnosed with colorectal polyps;
* Signing the written informed consent.

Exclusion Criteria:

* Patients with mental illness or severe functional disorder who cannot cooperate with colonoscopy;
* Patients with severe cardiopulmonary insufficiency;
* Patients with severe coagulation disorders or high bleeding risk (platelets <50×10⁹/L, INR >1.5; discontinuation of antithrombotic drugs should follow the 2012 Japanese Guidelines for Gastroenterological Endoscopy in Patients Undergoing Antithrombotic Treatment and the2017 Appendix on Anticoagulants Including Direct Oral Anticoagulants;
* Patients with severe electrolyte imbalances;
* Patients with acute peritonitis or suspected intestinal perforation;
* Patients with severe inflammatory bowel disease/toxic megacolon;
* Patients with polyposis syndromes (e.g., Peutz-Jeghers syndrome, Cronkhite-Canada syndrome, familial adenomatous polyposis [FAP], Lynch syndrome, etc.);
* Patients with stage 3 or higher hypertension (systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg);
* Patients with untreated severe abdominal hernia, intestinal obstruction, or advanced colorectal cancer;
* Patients with intestinal strictures of any cause;
* Cases requiring only endoscopic submucosal dissection (ESD);
* Pregnancy and lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
endoscopic diagnostic accuracy of polyps and adenomas | 1-7 days after polypectomy
  The overall proportion of correct classifications by endoscopy compared to the gold standard (pathology) in lesion level

SECONDARY OUTCOMES:
Modified high-risk adenoma (mHRA) detection rate | 1-7 days after polypectomy
  mHRA were defined with one of the following features:1. diameter ≥10 mm or 2. (tubulo)villous adenomas or 3. with high-grade dysplasia or 4. sessile serrated lesions (SSLs). SSLs were defined as lesions with at least one crypt showing a characteristic sessile serrated lesion-type appearance
Adenoma detection rate (ADR) | 1-7 days after polypectomy
  The number of participants with at least 1 adenoma divided by the total number of participants
Polyp detection rate (PDR) | 1-7 days after polypectomy
  The number of participants with at least 1 polyp divided by the total number of participants
Clinically relevant serrated polyp detection rate | 1-7 days after polypectomy
  Clinically relevant serrated polyps are defined as ≥10 mm serrated polyps (SPs, including hyperplastic polyps, SSLs, and traditional serrated adenomas) and >5 mm SPs in the proximal colon. Clinically relevant serrated polyp detection rate is defined as the number of participants with at least 1 clinically relevant serrated polyp divided by the total number of participants
early colorectal cancer detection rate | 1-7 days after polypectomy
  early colorectal cancer is defined as high-grade intraepithelial neoplasia or adenocarcinoma with submucosal invasion less than 1000μm (SM1)
the accuracy of the evaluation of invasion depth | 1-7 days after polypectomy
  The overall proportion of correct depth evaluation by endoscopy compared to the gold standard (pathology) in lesion level
the confidence of endoscopy diagnosis | during endoscopy diagnosis before polypectomy by the endoscopists
  the diagnostic confidence of the lession classification by the endoscopists
the accuracy of lession size evaluation | 1-7 days after polypectomy
  the proportion of correct estimated lession size by the endoscopists during examinaion with other endoscopists estimated by acquired images
The colonoscopy-relevant adverse events | 1-30 days after polypectomy
  aspiration pneumonia, perforation, bleeding, splenic injury/rupture, death, or others requiring hospitalization within 30 days after the colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguo Liu, M.D, Principal Investigator — Xijing Hospital of Digestive DIsease
Locations (1):
- Xijing Hospital of Digestive Disease, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No